CLINICAL TRIAL: NCT02693730
Title: Perceptions and Modulations of Visceral Sensations
Brief Title: Phenotyping IBS: Perceptions and Modulations of Visceral Sensations
Acronym: PMVS-P
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Emeran Mayer, MD, Professor and Director, University of California, Los Angeles
Other Study IDs: 2R01DK048351-15A1 (NIH); 2R01DK048351-15A1 (NIH)
Record Dates: First submitted 2016-01-12; First posted 2016-02-29 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Irritable Bowel Syndrome; Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Irritable Bowel Syndrome; IBS; Ulcerative Colitis; UC; Inflammatory Bowel Disease; IBD; Healthy Control; HC; Visceral Pain; Gut; Neuroimaging; fMRI; resting state; structural MRI; functional MRI; diffusion tensor imaging; MR Spectroscopy
MeSH Terms: conditions — Irritable Bowel Syndrome; Colitis, Ulcerative; Inflammatory Bowel Diseases; Visceral Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Stool samples will be collected from both IBS and IBD subjects. A full stool analysis will be performed on the stool of IBS subjects, whereas only calprotectin will be measured in the stool of IBD subjects.
  Blood will be collected from IBS subjects and HCs.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Healthy Control: Does not have diagnosis of irritable bowel syndrome (IBS) or inflammatory bowel disease (IBD) and is otherwise healthy and able to participate as defined by the exclusionary criteria.
- Irritable Bowel Syndrome (IBS): Diagnosed with IBS and meets the Rome III criteria, in the absence of red flag signs (i.e., unexplained weight loss, bloody stool, fever, anemia)
- Ulcerative Colitis (UC): Clinically and histologically confirmed diagnosis of ulcerative colitis

SUMMARY:
The purpose of this research study is to improve the understanding of irritable bowel syndrome (IBS) and its underlying cause. The investigators will use magnetic resonance imaging (MRI) to observe differences in the brain between people diagnosed with IBS compared to healthy controls and people with ulcerative colitis, a disease group that has already been characterized. By doing this correlative and comparative study, the investigators hope to gain knowledge on IBS in order to keep the field moving in the right direction and becoming one step closer to discovering effective treatments.

DETAILED DESCRIPTION:
Despite recent breakthroughs in research, irritable bowel syndrome (IBS) lacks a comprehensive mechanistic characterization. While the symptoms of this gastroenterological disorder have been described, the overall assessment of IBS has not led to sufficient treatment and management plans. By moving away from an over-reliance on a symptom-based approach and shifting towards a mechanism-based approach, investigators will be more knowledgeable as they attempt to address the disease. In order to accomplish this, the investigators will work with different patient subgroups, specifically IBS subjects, healthy controls (HCs), and disease control groups such as ulcerative colitis (UC). This will allow for the comparison of significant genetic, social, biological, and neurological findings between subgroups, which will help investigators grasp the differences present in people who suffer from IBS.

The investigators will approach the study in a couple different ways to characterize IBS in the best possible manner. Blood samples and MRI brain images will be collected so that the genetic and neurological factors associated with IBS can be explored. Given the highly interactive nature of the biological systems within the body, the investigators plan to explore the interaction between the brain and the immune system as well as the brain and the gut. In doing so, specific genes that contribute to IBS, as well as changes in the brain that contribute to or result from IBS, can be further scrutinized.Additionally, the immune system's influence on the brain in IBS patients can be compared to healthy controls or UC. All of this information will contribute to therapeutic studies in the future as investigators continue to develop both diagnostic tools and treatments for IBS patients.

Conducting this study necessitates the use of human subjects for research purposes. In total, the investigators will recruit 120 IBS subjects, 70 age-matched HCs, and 100 UC subjects. During the initial screening visit, the subject will complete a physical examination, a short psychological evaluation (MINI+), a pressure & heat sensitivity test, a quick blood draw, and a set of questionnaires. In total, this baseline visit will take roughly two hours.

On the second visit, the subject will return to complete more questionnaires and have their brains scanned by an MRI machine. The subject will then be disclosed of MRI safety procedures and once they are cleared, they will undergo a 60 minute scanning session with a certified MRI technician. Once this has been complete, the subject will have completed the study.

IBS female subjects that have indicated they would like to be part of the longitudinal study will return at 3 months, 6 months, 9 months, and 12 months for the same MRI procedure described above, with MR-Spectroscopy being an additional modality. They will also complete a 5 minute online survey every month for 9 months to assess their symptoms.

The Neuroimaging Core at the Center for Neurobiology of Stress will be responsible for all brain imaging analyses in years 4-5. Gene expression profiling assays and all microbiome related studies will occur at the Neuroscience Genomics Core Laboratory and the UCLA Center for Systems Biomedicine in years 4-5 as well.

ELIGIBILITY:
Inclusion Criteria for all IBS subjects:

* Meet Rome III criteria for IBS
* No red flag signs (i.e., weight loss, bloody stool, fever, anemia)

Inclusion Criteria for all UC subjects:

* Must have UC diagnosis that is clinically & histologically confirmed

Inclusion Criteria for all subjects:

* If woman of childbearing potential, must be willing to use contraception to avoid pregnancy during the course of the study
* If female, negative urine pregnancy tests at Screening & MRI Visit
* Willingness to participate in this study as evidenced by signed informed consent form
* ambulatory outpatient (does not depend on wheelchair for mobility)
* English is primary oral and written language

Exclusion Criteria for all subjects:

* Major medical intervention occurring in the next 6 months or in the past 6 months
* Presence of significant and ongoing medical problem interfering with participation
* Presence of major psychiatric diagnosis such as schizophrenia, bipolar disorder, PTSD, or Obsessive Compulsive disorder.
* Use of centrally acting medications that will interfere with neuroimaging testing (opiate analgesics, antidepressants).
* Left handed due to importance of laterality in neuroimaging
* Pregnancy or nursing
* Claustrophobia, Ferromagnetic Implants, or other problematic issues preventing subject participation in MRI
* Current or past history of chronic pain syndrome other than IBS in the IBS group
* History of gastrointestinal surgery other than uncomplicated appendectomy or cholecystectomy
* Use of investigational drugs, products, or devices within 28 days prior to screen and through study participation
* use of steroids in the last 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subject population will be made up of male and female adults between the ages of 18-60 and must fall into one of the following 3 groups: a) irritable bowel syndrome, b) ulcerative colitis, or c) healthy controls. Medical screening will be a physician or a nurse will confirm subject eligibility for the study.Subjects will be recruited from clinics and the community in and around Los Angeles Area.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2016-01; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Classifying patients with IBS and Ulcerative Colitis (UC) based on their brain "signatures" obtained from structural and functional MRI scanning. | MRI visit will be 45 min to 1 hour.
  Magnetic Resonance Imaging provides investigators with anatomical and functional images of the brain. Analytical neuroimaging tools demonstrate the unique brain properties of subjects in accordance with their conditions, referred to as brain "signatures."
Global and regional brain network alterations in IBS. | MRI visit will be 45 min to 1 hour.
  The architecture and wiring of the brain can be characterized using metrics describing the connectedness of brain regions, global and local network communication and signaling, and the contribution of each region to the network's structural integrity and information flow.
Possible biological mediators of observed IBS related brain network alterations | There will be a screening visit of about 1 hour with a single blood and stool sample; followed by about 40 minutes of on-line questionnaires.
  Proposed plausible pathophysiological mechanisms underlying structural and functional brain changes include: 1) Genetic and epigenetic factors; 2) neuroinflammation; 3) growth factor or stress-mediator induced neuroplastic changes; 4) microbiome derived metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Emeran Mayer, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Oppenheimer Center for Neurobiology of Stress and Resilience, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be stripped of identifiers before data sharing

REFERENCES:
- See also: Oppenheimer family center for Neurobiology of Stress at UCLA website — http://uclacns.org/